CLINICAL TRIAL: NCT06867653
Title: Different Re-training Durations in Basic Life Support Training Among Non-Professionals: A Three-Arm Randomized Controlled Trial
Brief Title: Different Re-training Durations in BLS Training Among Non-Professionals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 202007002RINB
Record Dates: First submitted 2025-02-12; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Education Curriculum
Keywords: retraining; basic life support

STUDY DESIGN:
Intervention Model Description: Three-armed randomized controlled Trial
Who Masked: Outcomes Assessor
Masking Description: During the skill assessment, two cameras recorded the process from different angles: one positioned from the feet towards the head of the manikin and the other from the left chest towards the right chest. Instructors, blinded to group allocation, later reviewed the recordings and assessed participants' performance using an evaluation form.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 45-minute retraining (Experimental): 45-minute retraining sessions
  Interventions: Other: Retraining
- 60-minute retraining (Experimental): 60-minute retraining sessions
  Interventions: Other: Retraining
- 75-minute retraining (Experimental): 75-minute retraining sessions
  Interventions: Other: Retraining

INTERVENTIONS:
Other: Retraining — Each retraining session begins with a 15-minute comprehensive review, followed by hands-on practice

SUMMARY:
Previous studies on compression-only CPR and AED training for the general public have primarily focused on the optimal retraining interval. However, the impact of different retraining durations remains unclear. This study explores how varying practice durations in Basic Life Support (BLS) training affect BLS performance among non-professionals.

DETAILED DESCRIPTION:
In this study, participants first underwent compression-only CPR and AED training. Before training, they completed a questionnaire on their perspectives on BLS retraining and basic demographic information. Knowledge tests, skill assessments, and attitude and confidence questionnaires were conducted both before and after training. During the skill assessment, two cameras recorded the process from different angles: one positioned from the feet towards the head of the manikin and the other from the left chest towards the right chest. Instructors, blinded to group allocation, later reviewed the recordings and assessed participants' performance using an evaluation form. Additionally, chest compressions were recorded using a computerized manikin (SkillReporter Resusci Anne®, Laerdal, Stavanger, Norway).

Participants were then randomly assigned to one of three groups based on different retraining durations:

1. 45-minute retraining sessions
2. 60-minute retraining sessions
3. 75-minute retraining sessions

All three groups underwent skill assessments and knowledge tests every three months before their respective retraining sessions. The retraining skill assessments followed the same procedure as the initial training. Each retraining session began with a 15-minute comprehensive review, followed by hands-on practice. Each participant practiced for approximately five minutes per cycle, which included two minutes of chest compressions, one minute of AED application, one minute of feedback, and one minute for role-switching. Based on this structure, participants in the 45-minute group completed two practice cycles, those in the 60-minute group completed three cycles, and those in the 75-minute group completed four cycles.

Both the initial training and retraining followed the American Heart Association (AHA) Heartsaver® CPR+AED course guidelines, with a participant-to-manikin ratio of 3:1 and a maximum of six participants per instructor. One year after the initial training, before the final skill assessment, participants completed the knowledge test and the attitude and confidence questionnaire. After the final skill assessment, they completed the CPR retraining perspectives questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years old

Exclusion Criteria:

* Subjects whose physical condition is unsuitable for the CPR training, such as those unable to squat, extend their arms fully, or individuals who are blind or deaf.
* Healthcare professionals and students majoring in healthcare-related fields.
* Individuals unwilling to sign the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Average compression rate | one year after the initial training
  The average compression rate during the skill assessment and the proportion of participants in each group with an average compression rate between 100-120 compressions per minute one year after the initial training

SECONDARY OUTCOMES:
Average compression depth | 3, 6, 9 and 12 months after the initial training
  The average compression depth and the proportion of participants in each group with an average compression depth between 5-6 cm during the skill assessment every three months
Average compression rate | 3 month, 6 months and 9 months after initial training
  The average compression rate and the proportion of participants in each group with an average compression rate between 100-120 compressions per minute at 3 month, 6 months and 9 months after initial training.
Chest recoil | 3, 6, 9 and 12 months after the initial training
  The proportion of complete chest recoil in each group every three months
Flow time | 3, 6, 9 and 12 months after the initial training
  The percentage of compression time over total assessment time in each group during the skill assessment
Correct hand placement | 3, 6, 9 and 12 months after the initial training
  The proportion of correct hand placement in each group during the skill assessment every three months
Pass rate | 3, 6, 9 and 12 months after the initial training
  The proportion of participants passing the assessment evaluated by instructors
Passing rates for each item | 3, 6, 9 and 12 months after the initial training
  The passing rate for each item on the evaluation form
Attitude | one year after the initial training
  The attitude questionnaire consists of two questions, each rated using a Likert scale, including 'strongly disagree,' 'disagree,' 'neutral,' 'agree,' and 'strongly agree.' When calculating the scores, 'strongly disagree' is assigned 1 point, 'disagree' 2 points, 'neutral' 3 points, 'agree' 4 points, and 'strongly agree' 5 points. A higher score indicates that participants place greater importance on the item.
Confidence | one year after the initial training
  The confidence questionnaire consists of three questions, each rated using a Likert scale, including 'strongly disagree,' 'disagree,' 'neutral,' 'agree,' and 'strongly agree.' When calculating the scores, 'strongly disagree' is assigned 1 point, 'disagree' 2 points, 'neutral' 3 points, 'agree' 4 points, and 'strongly agree' 5 points. A higher score indicates greater confidence.

OTHER OUTCOMES:
Perspectives questionnaire on retraining | one year after the initial training
  The perspective questionnaire on retraining consists of two questions: (1) How long do you think the interval for CPR retraining should be? (2) How long do you think the duration of a CPR retraining course should be? These two questions are open-ended.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Ju Hsieh, MD, PhD, Principal Investigator — National Taiwan University Hospital, Taipei, Taiwan
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan